CLINICAL TRIAL: NCT03866135
Title: The Relationship Between Bone Mineral Density, Disease Duration, and Activity in Patients With Ankylosing Spondylitis
Brief Title: Bone Mineral Density, Disease Duration, and Activity in Ankylosing Spondylitis
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Yaşar Keskin, Department of Physical Medicine and Rehabilitation, Principal Investigator, Medical Doctor, Bezmialem Vakif University
Other Study IDs: 11594
Record Dates: First submitted 2019-03-05; First posted 2019-03-07 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Ankylosing Spondylitis; Osteoporosis; BMD
MeSH Terms: conditions — Spondylitis, Ankylosing; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with osteoporosis: Osteoporosis has been operationally defined on the basis of bone mineral density (BMD) assessment. According to the WHO criteria, osteoporosis is defined as a BMD that lies 2.5 standard deviations or more below the average value for young healthy women (a T-score of <-2.5 SD)
- patients without osteoporosis: Bone mineral densities of patients were based on the World Health Organization (WHO) classification of a T score between -1 and -2.5 for osteopenia

SUMMARY:
Our clinical study aimed to evaluate the prevalence of osteoporosis (OP) in patients with ankylosing spondylitis (AS) and to investigate the relationship between clinical, disease activity, physical function and disease duration, and bone mineral density (BMD).

DETAILED DESCRIPTION:
In this cross-sectional study, patients who were admitted to the rheumatology clinic between 18 and 65 years of age and diagnosed as AS according to the modified New York diagnostic criteria were included

Patients group was divided two part as patients with (group 1)and without (group 2) osteoporosis.

The patient's global rating scale is a self-assessed scale of the patient with a grade of 10 (1: very bad, 5: moderate, 10: very good). To assess the disease activity, Bath ankylosing spondylitis disease index (BASDAI) and Bath ankylosing spondylitis functional index (BASFI) were evaluated. BASDAI is a self-assessment scale used to determine disease activity in patients with AS.

Schober measurement was used to evaluate lumbar mobility of the patients. Chest expansions were measured in all patients.

Body mass index (BMI) was calculated as kg/height m2. Erythrocyte sedimentation rate (ESH mm / h), C-reactive protein (CRP mg / l) levels were measured in all patients.

BMD measurements were made by using dual-energy x-ray absorptiometry (DEXA) and lumbar vertebra (L1-4) and left femur (femoral neck and total) regions. DEXA measurements (GE / LUNAR DPX PRO) were performed and the results were recorded using standard T score. Bone mineral densities of patients were based on the World Health Organization (WHO) classification of a T score between -1 and -2.5 for osteopenia; and a score of -2.5 for osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as AS according to the modified New York diagnostic criteria were included

Exclusion Criteria:

* Patients previously diagnosed with OP,
* Patients previously treated with OP,
* Patients with bone fractures previously associated with OP,
* Those using drugs that affect bone metabolism, metabolic bone diseases (Paget's -disease, osteomalacia, hyperparathyroidism),
* Diabetes mellitus,
* Hypothyroidism, hyperthyroidism,
* Patients with kidney, liver and intestinal diseases,
* Those using corticosteroids

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who were admitted to the rheumatology clinic between 25 and 65 years of age and diagnosed as AS according to the modified New York diagnostic criteria were included
Sampling Method: Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Bath ankylosing spondylitis disease index (BASDAI) | up to 6 month
  BASDAI, is a widely used patient-reported outcome to measure disease activity in AS. It comprises only six questions (Box 5.1).
  The answers to these questions are scored on a 0-10 NRS, which are anchored by 0 ("none") to 10 ("very severe"). The BASDAI sum score is calculated by the sum of questions 1-4 plus mean of questions 5 and 6, the total then divided by 5. The sum score ranges from 0 to 10, higher values indicate more active disease.
Bath ankylosing spondylitis functional index (BASFI) | up to 6 month
  Bath Ankylosing Spondylitis Functional Index (BASFI): this is the most frequently used tool to asses function in AS. It contains 10 questions on activities of daily living, which are scored with a rating scale from 0 (no functional impairments) to 10 (maximal impairment). The sum score ranges from 0 to 10, with higher values indicating worse functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No